CLINICAL TRIAL: NCT02623517
Title: A Novel Healthcare Information Technology Tool to Improve Care in Patients
Brief Title: A Novel Healthcare Information Technology Tool to Improve Care in Patients With Atrial Fibrillation
Acronym: AFCare
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Jonathan Hsu, Assistant Professor of Medicine, University of California, San Diego
Other Study IDs: 150702
Record Dates: First submitted 2015-12-01; First posted 2015-12-07 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
Keywords: CIED; AF; arrhythmia; atrial fibrillation; cardiac device; pacemaker; defibrillator
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Enrolled Subjects: The Enrolled Subjects group will comprise of 75 individuals who will be followed for 12 months for their atrial fibrillation condition. Data will be collected from subjects' devices for 12 months, and any needed changes or additions to therapy will be done. (ie: ablation, pacemaker setting changes, medication control).
- Registry Subjects: The Registry Subjects group will comprise of screened patients who do not exhibit symptoms of atrial fibrillation at the time of screening. The already collected data from the patient's device during the screening visit will be kept and put into a registry.

SUMMARY:
Patients with implantable heart devices including pacemakers, defibrillators, and cardiac monitors may not seek regular medical care related to their implanted devices. These devices are capable of detecting abnormal heart rhythms or other device abnormalities that may benefit from clinical action or oversight. A novel healthcare information technology has been developed and is being implemented clinically for screening of patients with cardiac rhythm devices who seek care in the emergency room setting. This study seeks to examine differences in detection of cardiac rhythm disturbances including atrial fibrillation (AF) with utilization of this new screening technology, and how often treatment plans change in patients who have a heart rhythm abnormality detected.

DETAILED DESCRIPTION:
This study is a prospective, observational study designed to evaluate the use of the Geneva Healthcare Patient Population Management platform to detect AF (atrial fibrillation) in patients with CIEDs (cardiovascular implantable electronic devices) in the emergency room setting, and assess the feasibility of sub-specialty cardiac electrophysiology (EP) care of these patients. This is a PI-initiated study and there are currently no plans to conduct this study at any other sites.

The investigators plan to use the Geneva Healthcare Patient Population Management platform to detect AF in patients with CIEDs and will utilize a clinical excellence team of nurse practitioners and research assistants to ensure that appropriate treatment of AF is pursued. UCSD (University of California, San Diego) has used the Geneva Patient Population Management Platform for clinical purposes since September, 2012 at both emergency room sites at Hillcrest and Thornton. The platform is not an experimental device.

After the patient's device is interrogated in the usual fashion by placing a wand over the patient, with downloading of information to each device manufacturers interrogator, the information is uploaded to the Geneva platform, where it is organized for a physician to interpret. After the data has been processed and organized on the password protected system, the data retrieved from the CIED will be uploaded to UCSD's electronic medical record system, EPIC, by the hospital personnel. For the purposes of this study, the Geneva Healthcare PPM (Patient Population Management) platform is simply a tool used to collect relevant device data in the ER setting.

The investigators plan to clinically screen all patients who are evaluated in either of two UCSD emergency departments who have any cardiac rhythm device. This ER screening will be incorporated into standard clinical practice and will be conducted by EP staff. The goal will be to detect all patients with AF and to refer them for direct electrophysiology evaluation. Patients with AF will have data captured from physiologic and arrhythmia data collected by the Geneva Healthcare PPM platform from the point-of-care interrogation in the ER (emergency room) or by home monitoring.

A Clinical Excellence Team of physicians, nurse practitioners, and nurses will direct identified patients with AF to appropriate treatment by referral to an EP subspecialist for treatment considerations including rate control, rhythm control, stroke prophylaxis therapy, and ablation therapy. The patient will be offered a clinic appointment with an EP subspecialist. Patients who have been identified with atrial fibrillation will be referred to research staff. If the patient is interested in participation in the main trial, informed consent will be obtained by one of the study investigators or research coordinators. Patients who are enrolled in the trial will be followed through their course of standard clinical treatment for atrial fibrillation for 12 months, including both ablation and medication therapy. Outcomes including morbidity, mortality, hospitalization, healthcare utilization, and recurrent AF will be evaluated in all patients (including those who are taken to ablation vs. those who are not). If a patient refuses to be referred to an EP subspecialist, the patient will not be approached for research. The patient will be encouraged to follow-up with any previous physician they have recently seen, including a primary care physician and/or cardiologist for standard clinical care.

The investigators propose a pilot clinical excellence study leveraging innovative healthcare information technology tools to capture patients with AF and CIEDs, and efficiently route these patients for guideline-based treatment with a goal for appropriate radiofrequency catheter ablation of AF and/or medical therapy. The investigators' mission is to evaluate the ability to detect AF in patients with cardiac rhythm devices with this novel healthcare technology, increase access to proper medical and procedural therapy for AF, and evaluate a centralized repository for follow-up of clinical results and outcomes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Atrial Fibrillation
* Patients presented in the UCSD E.D with a CIED
* Patient willingness to participate

Exclusion Criteria:

* Any medical condition that may prevent patient's ability to participate
* No indication of Atrial Fibrillation
* Patient unable to follow-up at UCSD or follow research instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiovascular implantable electronic devices (CIED), including pacemakers, defibrillators, and cardiac resynchronization therapy devices
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-05; Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of atrial fibrillation in patients with CIEDs | two years
  To establish the prevalence of device detected atrial tachyarrhythmia episodes (most commonly AF) in patients who have device interrogations performed in the Emergency Room by the Geneva Healthcare Patient Population Management Platform
The prevalence of cardiac electrophysiology referrals from the E.D | two years
  To establish the prevalence of cardiac electrophysiology referral in a population of patients with cardiac rhythm devices but no Geneva Healthcare Patient Population Management Platform routine interrogation versus routine interrogation in the emergency room.
The patient population with AF that are treated with catheter ablation | two years
The patient population with AF that are treated with rate-control therapy | two years
The patient population with AF that are treated with rhythm control drug therapy | two years
The patient population with AF that are treated with oral anticoagulation for stroke prophylaxis | two years
The prevalence of device and lead malfunctions in patients with CIEDs. | two years
  To investigate the prevalence of device and lead malfunction in a population of patients with cardiac rhythm devices undergoing interrogation by the Geneva Healthcare Patient Population Management Platform.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Hsu, MD, Principal Investigator — UC San Diego School of Medicine; Sulpizio Cardiovascular Center
Locations (1):
- Sulpizio Cardiovascular Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lloyd-Jones DM, Wang TJ, Leip EP, Larson MG, Levy D, Vasan RS, D'Agostino RB, Massaro JM, Beiser A, Wolf PA, Benjamin EJ. Lifetime risk for development of atrial fibrillation: the Framingham Heart Study. Circulation. 2004 Aug 31;110(9):1042-6. doi: 10.1161/01.CIR.0000140263.20897.42. Epub 2004 Aug 16. PMID 15313941
- [Result] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Result] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222
- [Result] Glotzer TV, Daoud EG, Wyse DG, Singer DE, Ezekowitz MD, Hilker C, Miller C, Qi D, Ziegler PD. The relationship between daily atrial tachyarrhythmia burden from implantable device diagnostics and stroke risk: the TRENDS study. Circ Arrhythm Electrophysiol. 2009 Oct;2(5):474-80. doi: 10.1161/CIRCEP.109.849638. Epub 2009 Aug 4. PMID 19843914
- [Result] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D; Heart Rhythm Society Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. 2012 HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design: a report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. Developed in partnership with the European Heart Rhythm Association (EHRA), a registered branch of the European Society of Cardiology (ESC) and the European Cardiac Arrhythmia Society (ECAS); and in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), the Asia Pacific Heart Rhythm Society (APHRS), and the Society of Thoracic Surgeons (STS). Endorsed by the governing bodies of the American College of Cardiology Foundation, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, the Asia Pacific Heart Rhythm Society, and the Heart Rhythm Society. Heart Rhythm. 2012 Apr;9(4):632-696.e21. doi: 10.1016/j.hrthm.2011.12.016. Epub 2012 Mar 1. No abstract available. PMID 22386883